CLINICAL TRIAL: NCT00608907
Title: An Open-Label Study to Assess the Effect of CYP3A4 Induction on the Pharmacokinetics of VELCADE (Bortezomib)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-CAN-1006
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Myeloma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Bortezomib; Rifampin; Dexamethasone

ARMS (3):
- VELCADE (Experimental): Control arm, bortezomib 1.3 mg/m^2 on days 1, 4, 8, 11 over a 21-day treatment cycle.
  Interventions: Drug: bortezomib
- VELCADE + rifampicin (Experimental): Treatment Arm, bortezomib 1.3 mg/m^2 on days 1, 4, 8, 11 over a 21-day treatment cycle, rifampicin 600 mg once daily days 4 to 10 in cycle 3.
  Interventions: Drug: bortezomib, rifampicin
- VELCADE + dexamethasone (Experimental): Treatment arm, bortezomib 1.3 mg/m^2 on days 1, 4, 8, 11 over a 21-day treatment cycle, dexamethasone 40 mg once daily days 1 to 4, and 9 to 12 in cycle 3.
  Interventions: Drug: bortezomib, dexamethasone

INTERVENTIONS:
Drug: bortezomib — 1.3 mg/m^3 on days 1, 4, 8, 11 over a 21-day treatment cycle
  Other Names: VELCADE
  Arms: VELCADE
Drug: bortezomib, rifampicin — bortezomib 1.3 mg/m^2 on days 1, 4, 8, 11 over a 21-day treatment cycle, rifampicin 600 mg once daily days 4 to 10 in cycle 3
  Other Names: bortezomib; rifampicin
  Arms: VELCADE + rifampicin
Drug: bortezomib, dexamethasone — bortezomib 1.3 mg/m^2 on days 1, 4, 8, 11 over a 21-day treatment cycle, dexamethasone 40 mg once daily days 1 to 4, and 9 to 12 in cycle 3
  Other Names: bortezomib; dexamethasone
  Arms: VELCADE + dexamethasone

SUMMARY:
The primary purpose of this Phase I study is to evaluate the effect of the co-administration of CYP3A4 inducers on the pharmacokinetics profile of VELCADE (bortezomib). Rifampicin will be used to assess the effect of a strong CYP3A4 inducer and dexamethasone to assess the effect of a relatively weak inducer. This study is also to evaluate the impact of CYP3A4 inducers on the pharmacodynamics (PD) of VELCADE and the safety profile of VELCADE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 18 years of age.
* Has documented relapsed or refractory multiple myeloma or NHL following prior anti-neoplastic treatment.
* Female patients must be post menopausal for at least 1 year (must not have had a natural menses for at least 12 months), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; have a negative serum β-HCG or a negative urine pregnancy test at screening. (an alternative to oral contraceptives should be used if the patient is randomized to Arm B with rifampicin).
* Male patients must agree to use an acceptable method of contraception (for themselves or female partners as listed above) for the duration of the study.
* Must be able to swallow capsules/tablets whole (without chewing, crushing, or opening).
* Agree to refrain from the use of any methylxanthine-containing products, including caffeine (e.g., chocolate bars or beverages, coffee, teas, or colas), on Day 11 of Cycles 2 and 3.
* Agree to refrain from the use of any products containing nicotine, alcohol, quinine, grapefruit juice, or Seville oranges from 7 days before the first administration of VELCADE through completion of the 72-hour PK blood sample collection (post Day 11 VELCADE dose) in Cycle 3.

Exclusion Criteria:

* Diagnosis or treatment of a malignancy other than multiple myeloma or NHL within 1 year of randomization, or who have previously been diagnosed with a malignancy other than multiple myeloma or NHL and have any radiographic or biochemical marker evidence of malignancy.
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, psychiatric, or metabolic disturbances.
* Known or suspected hypersensitivity or intolerance to rifampicin and/or other antibiotics, corticosteroids, boron or mannitol.
* Peripheral neuropathy or neuropathic pain Grade 2 or higher.
* Preplanned surgery or procedures that would interfere with the conduct of the study or major surgery within 2 weeks before randomization.
* History of disallowed therapies:

  * Prior treatment with VELCADE.
  * Any drugs or agents that inhibit (e.g., cimetidine, erythromycin, fluoxetine, ketoconazole, paroxetine) or induce (e.g., carbamazepine, glucocorticoids, phenobarbital, phenytoin, St. John's Wort) CYP2C19 or CYP3A4 within 28 days before the first administration of VELCADE.
  * Any exposure to rifampicin or corticosteroids within 28 days of screening.
  * Have received an investigational agent or used an investigational medical device within 28 days before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study.
* Female patient who is pregnant or breastfeeding.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (9):
- Hematology Institute - Davidoff Center - Rabin Medical Center, Petah Tikva, Israel
- Divisione di Ematologia - Ospedale S Eugenio - P. le dell'Umanesimo, Rome, Italy
- Poland (2):
  - Medical Academy - Dept of Hematology and Transplantology, Gdansk
  - Klinika Nowotworow Ukladu - Chlonnego - Centrum Onkologii - Instytut, Warsaw
- South Africa (3):
  - Hematological Oncology, Parow, Cape Town
  - Department of Hematology - University of the Free State, Bloemfontein
  - Department of Medical Oncology - Ward 51 - Pretoria Academic Hospital, Pretoria
- United Kingdom (2):
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Derriford, Plymouth
  - Hematology Department Combined Laboratories - Derriford Hospital, Plymouth

RESULTS

PARTICIPANT FLOW:
Groups:
- VELCADE: Control arm, bortezomib 1.3 mg/m^2 IV bolus on days 1, 4, 8, 11 over a 21-day treatment cycle.
- VELCADE + Rifampicin: Treatment Arm, bortezomib 1.3 mg/m^2 IV bolus on days 1, 4, 8, 11 over a 21-day treatment cycle, rifampicin 600 mg oral tablet once daily days 4 to 10 in cycle 3.
- VELCADE + Dexamethasone: Treatment arm, bortezomib 1.3 mg/m^2 IV bolus on days 1, 4, 8, 11 over a 21-day treatment cycle, dexamethasone 40 mg oral tablet once daily days 1 to 4, and 9 to 12 in cycle 3.
Period: Overall Study
Arm/Group | VELCADE | VELCADE + Rifampicin | VELCADE + Dexamethasone
Started | 30 | 13 | 18
Completed | 18 | 13 | 17
Not Completed | 12 | 0 | 1
Not completed — Adverse Event | 6 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VELCADE | VELCADE + Rifampicin | VELCADE + Dexamethasone | Total
Number analyzed (Participants) | 30 | 13 | 18 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 8 | 8 | 30
  >=65 years | 16 | 5 | 10 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.86) | 60.2 (9.97) | 62.3 (11.72) | 63.0 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 9 | 31
  Male | 15 | 6 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) 0-72 Hours
Time Frame: Cycle 3 day 14 (72 hours post last dose)
Population: Pharmacokinetic (PK) evaluable population, include all subjects completed 3 cycles of treatment and all PK assessments during the first 3 cycles of the study.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | VELCADE + Rifampicin | VELCADE + Dexamethasone | VELCADE
Number analyzed (Participants) | 6 | 7 | 12
ng*h/mL | 123 (34.2) [48.14 to 63.06] | 170 (64.5) [82.28 to 105.21] | 215 (58.4)

ADVERSE EVENTS:
Arm/Group | VELCADE | VELCADE + Rifampicin | VELCADE + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 14/30 | 5/13 | 7/18
Other Adverse Events (participants affected / at risk) | 28/30 | 13/13 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE (N=30) | VELCADE + Rifampicin (N=13) | VELCADE + Dexamethasone (N=18)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Catheter Site Haemorrhage (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Disease Progression (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Thrombosis in Device (General disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 1
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Meningitis Listeria (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Paralysis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Circulatory Collapse (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE (N=30) | VELCADE + Rifampicin (N=13) | VELCADE + Dexamethasone (N=18)
Anaemia (Blood and lymphatic system disorders) | 7 | 3 | 6
Neutropenia (Blood and lymphatic system disorders) | 7 | 6 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 5 | 8
Blepharitis (Eye disorders) | 1 | 0 | 2
Conjunctivitis (Eye disorders) | 4 | 3 | 1
Eye pain (Eye disorders) | 3 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 3
Abdominal Distension (Gastrointestinal disorders) | 4 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 8 | 6 | 3
Chills (General disorders) | 4 | 2 | 1
Oedema Peripheral (General disorders) | 8 | 1 | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 2 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 2
Herpes Zoster (Infections and infestations) | 4 | 1 | 2
Influenza (Infections and infestations) | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0
Oral Herpes (Infections and infestations) | 1 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 2 | 7
Rib Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Weight Decreased (Investigations) | 2 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 1 | 0
Enzyme Abnormality (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 4
Dizziness (Nervous system disorders) | 5 | 5 | 2
Dysgeusia (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 11 | 3 | 4
Neuralgia (Nervous system disorders) | 3 | 3 | 6
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 2 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 6 | 10
Dysthymic Disorder (Psychiatric disorders) | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 1 | 2
Nightmare (Psychiatric disorders) | 2 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 3 | 2 | 2
Testicular Pain (Reproductive system and breast disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 4
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hypertension (Vascular disorders) | 1 | 1 | 3
Dry Eye (Eye disorders) | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 11 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No